CLINICAL TRIAL: NCT05005741
Title: A Randomized Controlled, Open-label, Multi-center Study With 16-week Beinaglutide or Dulaglutide Assessing Effects on Glucose Control and Weight Loss in Type 2 Diabetes With Overweight or Obesity.
Brief Title: The Effects of Glucose Control and Weight Loss Between Beinaglutide and Dulaglutide in Type 2 Diabetes With Overweight or Obesity.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhiguang Zhou, Director of The National Clinical Research Center for Metabolic Diseases, and Key Laboratory of Diabetes Immunology, Ministry of Education, and Department of Endocrinology, The Second Xiangya Hospital of Central South University., Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BENEFIT 1
Record Dates: First submitted 2021-08-09; First posted 2021-08-13 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2; Overweight or Obesity
Keywords: GLP-1 receptor agonist; Beinaglutide; Dulaglutide; Type 2 diabetes; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity | interventions — glucagon-like peptide 1 (7-36); dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beinaglutide (Experimental)
  Interventions: Drug: Beinaglutide
- Dulaglutide (Active Comparator)
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: Beinaglutide — Patients received beinaglutide subcutaneously three times a day for 16 weeks, the dose of beinaglutide escalate from 0.06mg to 0.2mg per 3-7 days according to subject's specific situation.
  Other Names: GLP-1 receptor agonist
  Arms: Beinaglutide
Drug: Dulaglutide — Patients received 1.5mg Dulaglutide subcutaneously once-weekly for 16 weeks.
  Other Names: Trulicity; GLP-1 receptor agonist
  Arms: Dulaglutide

SUMMARY:
This study is a multi-center, open label, randomized controlled trial that main purpose of this study is to evaluate the differences of glucose control and weight loss between Beinaglutide and Dulaglutide in type 2 diabetes with overweight or or Obesity.

DETAILED DESCRIPTION:
About 2/3 of patients with type 2 diabetes are overweight or obese in China, several studies had confirmed that overweight and obesity could cause type 2 diabetes. GLP-1 receptor agonist could control diabetes meanwhile loss the patient weight. This is a multi-center, openlabel, 1:1 randomized controlled trial to investigate the differences of glucose control and weight loss between two GLP-1 receptor agonist, Beinaglutide and Dulaglutide, in type 2 diabetes with overweight or Obesity. The study comprises the 0-2 weeks of screening period and the 16-week intervention period. 120 patients according to the inclusion/exclusion criteria would recruit from 4 sites in China, then the participant will be randomized to three times a day of subcutaneous beinaglutide(dose escalate to 0.2mg), or once-weekly of 1.5mg subcutaneous dulaglutide for 16-week. The primary endpoint is the change from baseline to week 16 in HbA1c. The second endpoint is the change from baseline to week 16 in weight.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 70 years old from all sex;
2. Diagnosed with type 2 diabetes and HbA1c between 7% to 10%;
3. BMI from 24 to 35kg/m² or waistline longger than 90cm（male）/85cm（female）;
4. Volunteer to participate in the study with informed consent;

Exclusion Criteria:

1. Type 1 diabetes or other specific types of diabetes;
2. Taking drugs of GLP-1 receptor agonist、TZDs and SGLT2 inhibitor within 3 months of screening;
3. Taking insulin or insulin analogues more than 7 days within 3 months of screening;
4. Pregnancy, breastfeeding or planned pregnancy;
5. History of acute or chronic pancreatitis;
6. Taking glucocorticoids(oral or intravenous) continuously more than 7 days within 6 months of screening;
7. Alanine aminotransferase or aspartate transaminase more than 3 times of the normal upper limit, total bilirubin more than 2 times of the normal upper limit;
8. renal impairment (estimated glomerular filtration rate<60mL/min per 1.73 m²);
9. History of gastrointestinal disease;
10. History of malignant tumor within 5 years of screening;
11. History of organ transplantation or AIDS;
12. History of glaucoma;
13. History of hyperthyroidism or hypothyroidism;
14. History of medullary thyroid carcinoma or multiple endocrine neoplasia II;
15. History of abnormal of Calcitonin or thyroid tumor;
16. History of alcohol abuse;
17. Recruited by other clinical trials within 3 months of screening;
18. Taking drugs of weight loss within 3 months of screening;
19. History of bariatric surgery;
20. History of mental disorders;
21. History of rheumatic diseases or autoimmune diseases;
22. Allergic to beinaglutide or dulaglutide;
23. Participants who estimated would not be suitable for the study by the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
haemoglobin A1c(HbA1c) | From baseline to 16 week.
  Absolute changes from baseline in HbA1c at week 16.

SECONDARY OUTCOMES:
Weight loss | From baseline to 16 week.
  The proportion of weight loss from baseline to week 16；the proportion of subjects who loss 5% weight at week 16 compares baseline.
GLucose | From baseline to 16 week.
  Absolute changes from baseline in fasting glucose and postprandial glucose at week 16.
Body Mass Index(BMI) | From baseline to 16 week.
  Absolute changes from baseline in BMI in at week 16, body mass index (BMI) was calculated as the body weight (kg)/height (m)2.
Waistline | From baseline to 16 week.
  Absolute changes from baseline in waistline at week 16.
Hipline | From baseline to 16 week.
  Absolute changes from baseline in hipline at week 16.
Serum total cholesterol | From baseline to 16 week.
  Absolute changes from baseline in serum total cholesterol at week 16.
Serum triglycerides | From baseline to 16 week.
  Absolute changes from baseline in triglycerides at week 16.
Serum Low Density Lipoprotein-Cholesterol(LDL-C) | From baseline to 16 week.
  Absolute changes from baseline in LDL-C at week 16.
Serum High Density Lipoprotein-Cholesterol(HDL-C) | From baseline to 16 week.
  Absolute changes from baseline in HDL-C at week 16.
Adipose tissue of liver | From baseline to 16 week.
  Absolute changes from baseline in HDL-C at week 16, adipose tissue of liver will be mersured by Fibroscan, a device useing an ultrasound transducer probe to vibrations of liver presenting adipose tissue content.
Homeostasis model assessment for insulin resistance(HOMA-IR) | From baseline to 16 week.
  Absolute changes from baseline in HOMA-IR at week 16, HOMA-IR was calculated as [fasting glucose (mmol/L)× fasting insulin (μU/ml)/22.5].
Homeostasis model assessment for β cell(HOMA-β) | From baseline to 16 week.
  Absolute changes from baseline in HOMA-β at week 16, HOMA-β was calculated as [20× fasting insulin (μU/ml)/fasting glucose (mmol/L)-3.5].

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No